CLINICAL TRIAL: NCT04584372
Title: Effects of Dietary Nitrate on Vascular Function, Blood Pressure, the Oral Microbiome, and Biomarkers of Systemic Inflammation in Hypertensive Older Adults: a Randomized, Placebo-controlled Crossover Study
Brief Title: Dietary Nitrate, Vascular Function and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vienna (Other)
Collaborators: Medical University of Vienna (Other); Queensland University of Technology (Other); Flinders University (Other); Edith Cowan University (Other)
Responsible Party: Principal Investigator, Oliver Neubauer, Dr PhD, PD, University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UVienna_Dietary nitrate
Record Dates: First submitted 2020-09-29; First posted 2020-10-14 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Hypertension; Inflammation
Keywords: dietary nitrate; inorganic nitrate-nitrite-nitric oxide pathway; oral microbiome; chronic low-grade inflammation; vascular integrity; high blood pressure; cardiovascular health
MeSH Terms: conditions — Hypertension; Inflammation

STUDY DESIGN:
Intervention Model Description: Prospective, mono-center, randomized, double-blind, placebo-controlled, crossover study
  The study will involve a randomized, placebo-controlled crossover design, with two 4-week treatment periods separated by a 4-week washout period. The two treatments will consist of a 4-week high-nitrate (HI-NI) and a 4-week low-nitrate (LO-NI, i.e., placebo) intervention in older adults with treated grade 1 hypertension, on the background of a low-nitrate diet and unaltered lifestyle.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The two treatment arm will consist of a 4-week high-nitrate (HI-NI) intervention (using nitrate-rich beetroot juice) and a 4-week low-nitrate (LO-NI) intervention using nitrate-depleted beetroot juice as the placebo. All products will be obtained from the same supplier (James White Drinks Ltd., UK). The nitrate-depleted beetroot juice is generated for research purposes only. The two juices will be indistinguishable by taste, color, smell and packaging. The investigators involved in the data acquisition and analysis will be blind to the trial allocation until the study has been completed and all analyses have been performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-nitrate (HI-NI) intervention (Active Comparator): The 'active treatment' arm will involve daily consumption of 2×70 mL nitrate-rich (HI-NI) beetroot juice (70 mL with breakfast and 70 mL with dinner) over an intervention period of 4 weeks.
  Interventions: Dietary Supplement: High-nitrate intervention
- Low-nitrate (LO-NI) intervention (Placebo Comparator): The placebo treatment arm daily consumption of 2×70 mL nitrate-depleted (LO-NI) beetroot juice (70 mL with breakfast and 70 mL with dinner) an intervention period of 4 weeks.
  Interventions: Dietary Supplement: Low-nitrate intervention

INTERVENTIONS:
Dietary Supplement: High-nitrate intervention — The 2×70 mL of nitrate-rich (i.e., 'high nitrate') beetroot juice contains 12.9 mmol nitrate (NO3-).
  Other Names: HI-NI
  Arms: High-nitrate (HI-NI) intervention
Dietary Supplement: Low-nitrate intervention — The 2×70 mL of nitrate-depleted (i.e., 'low nitrate') beetroot juice contains 0.04 mmol (or less) nitrate.
  Other Names: LO-NI
  Arms: Low-nitrate (LO-NI) intervention

SUMMARY:
The risk for cardiovascular diseases (CVD) increases with advancing age. Developing effective lifestyle-based strategies to promote, preserve or restore cardiovascular health with aging is a high priority. The overall aim of this clinical research is to investigate the innovative concept that an increased intake of dietary nitrate (through beetroot juice) could be a feasible adjuvant therapy to treat elevated blood pressure and improve blood vessel function in older adults.

Inorganic dietary nitrate, found in beetroot and green leafy vegetables, is a source of nitric oxide (NO), a signaling molecule that is important for cardiovascular health. NO is also produced in the human body, but the body's production and availability of NO decrease during ageing and CVD. The declined NO availability is associated with impaired blood vessel function, unresolved inflammatory responses, and an increased CVD risk. Dietary nitrate is an additional NO source. Following the intake of nitrate, NO is produced in a pathway that involves commensal bacteria in the mouth. So far, little is known about whether dietary nitrate improves cardiovascular health in older populations with high blood pressure.

The aim of this randomized, placebo-controlled crossover study is to investigate whether the daily intake of nitrate-rich beetroot juice over four weeks translates into improved cardiovascular health-related outcomes in older adults with treated mild high blood pressure. Men and women, between the ages of 55 and 70 years, who have been diagnosed with grade 1 high blood pressure and who are taking two or more blood-pressure lowering medications will be recruited. The study will investigate whether the increased dietary nitrate intake further lowers blood pressure and improves blood vessel function. A specific aim is to examine whether the nitrate intake results in favorable changes in the oral bacteria community and the systemic inflammatory status, and whether these changes correlate with cardiovascular-related outcomes. This research will offer information on the value of dietary nitrate to counteract chronic inflammation, the latter of which plays a role in developing or worsening cardiovascular disorders, such as high blood pressure.

The expected results of this study will provide important new evidence of whether nitrate-rich beetroot juice could be a key component of therapeutic interventions to improve cardiovascular health in individuals with high blood pressure.

DETAILED DESCRIPTION:
This clinical research is funded by the Austrian Science Fund (FWF, project number: KLI 858). It is based on close collaborations between the University of Vienna and the Medical University of Vienna, with the Department of Clinical Pharmacology at the Medical University of Vienna as the clinical trial center and Prof. M.D. Michael Wolzt as the trial center's coordinating physician. The sponsor is the University of Vienna, as represented by the Principal Investigator Dr. Oliver Neubauer (Research Platform Active Ageing). International collaborations include Dr. Catherine Bondonno, Prof. Hodgson (both Edith Cowan University) Dr. Jonathan Peake (Queensland University of Technology), and Prof. Richard Woodman (Flinders University) (all Australia).

Wider research context / theoretical framework:

Aging is a major risk factor for cardiovascular disease (CVD). Developing effective strategies to improve cardiovascular health with ageing is a high priority. Emerging data indicate that inorganic dietary nitrate, found in green leafy vegetables and beetroot juice (BRJ), is important for cardiovascular health (Blekkenhorst et al. 2018). These data suggest that small increases in nitrate intake among those with elevated risk for CVD would have a substantial impact, by improving the bioavailability of nitric oxide (NO) through the enterosalivary nitrate- nitrite-NO pathway (involving the oral microbiome). Results from the study group's research suggest beneficial short-term effects of nitrate-rich BRJ on blood pressure and vascular inflammation markers in healthy older adults (Raubenheimer et al. 2017).

Hypotheses / research questions / objectives:

The proposed clinical study is aimed to examine whether the daily consumption of 2×70 mL BRJ over 4 weeks translates into improved clinical outcomes in older adults with treated grade 1 hypertension. The primary hypothesis is that the increased dietary nitrate intake lowers blood pressure and improves vascular function. The secondary hypotheses are that the increased dietary nitrate intake results in changes in the oral microbiome, favorably modulates the systemic inflammatory status, and that these changes correlate with cardiovascular-related outcomes.

Approach / methods:

This randomized, placebo-controlled crossover study will involve two 4-week treatment periods, consisting of interventions with nitrate-rich BRJ and nitrate-depleted BRJ, separated by a 4-week washout period. Thirty-five men and women, between the ages of 55 and 70 years, who have been diagnosed with grade 1 hypertension will be recruited. Twenty-nine participants will be required to complete the study, based on power/sample size calculations with the forearm blood flow (FBF) response to acetylcholine and 24 h-ambulatory systolic blood pressure as the primary endpoints. Principal secondary endpoints are the number of CD11b-expressing blood granulocytes and the FBF response to glyceryltrinitrate. Among various additional secondary and exploratory endpoints, plasma nitrate and nitrite and a broad range of inflammation biomarkers will be measured. Furthermore, the oral microbiome will be analyzed.

Level of originality / innovation:

Beneficial effects of nitrate have predominantly been observed in healthy populations, but evidence of cardiovascular benefits and anti-inflammatory effects in clinical populations is limited (Raubenheimer et al. 2019). This study addresses the need to determine the efficacy of dietary nitrate to improve cardiovascular health and counteract chronic low-grade inflammation in humans at risk of CVD.

ELIGIBILITY:
Inclusion Criteria:

* Ambulant male and females between 55 and 75 years of age, inclusive
* Resting systolic blood pressure between 130 and 170 mmHg, inclusive
* Written informed consent

Exclusion Criteria:

* Diastolic blood pressure >110 mmHg
* Type 1 or 2 diabetes mellitus or fasting glucose >7.0 mmol/L
* Any evidence of acute or chronic disease such as symptomatic cardiovascular or peripheral vascular disease, moderate or severe chronic kidney disease (estimated glomerular filtration rate (GFR) <50 ml/min)), or cancer which is not in remission
* Consumption of ≥5 serves of vegetables per day
* Consumption of a diet estimated to contain >200 mg/d of nitrate
* Being vegan or vegetarian
* BMI ≥35 kg/m2 or <18.5 kg/m2
* Use of nitric oxide donors, organic nitrites/nitrates, sildenafil and related drugs, anti-coagulation, non-steroidal anti-inflammatory or statin-related drugs
* Use of antibacterial mouthwash (volunteers willing to cease using antibacterial mouth wash for a period of 4 weeks before randomisation will be included)
* Use of antibiotics (within previous 2 months)
* A change in drug therapy likely to influence blood pressure or major secondary outcomes within the previous month, or the likelihood that drug therapy would change during the study
* Current or recent (within previous 3 months) engagement in regular structured exercise training (more than 2 hours of moderate to more intense exercise per week)
* Current or recent (within previous 6 months) loss or gain of >6% of body weight
* Current or recent (<12 months) regular smoking of >5 cigarettes/day
* Alcohol intake >140 g per week for women or >210 g per week for men and/or binge drinking behaviour
* Inability or unwillingness to follow the study protocol
* Pregnancy or lactation

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Change in forearm blood flow (FBF) response to acetylcholine | Change from baseline FBF at 4 weeks of the HI-NI intervention
  Vascular function
Change in forearm blood flow (FBF) response to acetylcholine | Change from baseline FBF at 4 weeks of the LO-NI intervention
  Vascular function
Change in 24 hour-ambulatory systolic blood pressure | Change from baseline 24 hour-ambulatory systolic blood pressure at 4 weeks of the HI-NI intervention
  Blood pressure
Change in 24 hour-ambulatory systolic blood pressure | Change from baseline 24 hour-ambulatory systolic blood pressure at 4 weeks of the LO-NI intervention
  Blood pressure

SECONDARY OUTCOMES:
Change in granulocyte CD11b expression | Change from baseline granulocyte CD11b expression at 4 weeks of the HI-NI intervention
  Vascular inflammation biomarker
Change in granulocyte CD11b expression | Change from baseline granulocyte CD11b expression at 4 weeks of the LO-NI intervention
  Vascular inflammation biomarker
Change in forearm blood flow (FBF) response to glyceryltrinitrate | Change from baseline FBF at 4 weeks of the HI-NI intervention
  Vascular function
Change in forearm blood flow (FBF) response to glyceryltrinitrate | Change from baseline FBF at 4 weeks of the LO-NI intervention
  Vascular function

OTHER OUTCOMES:
Change in clinical blood pressure | Change from baseline clinical blood pressure at 4 weeks of the HI-NI intervention
  Blood pressure
Change in clinical blood pressure | Change from baseline clinical blood pressure at 4 weeks of the LO-NI intervention
  Blood pressure
Change in plasma nitrate and nitrite | Change from baseline plasma nitrate and nitrite at 4 weeks of the HI-NI intervention
  Marker for nitrate bioavailability and functioning of the enterosalivary nitrate-nitrite-nitric oxide (NO) pathway
Change in plasma nitrate and nitrite | Change from baseline plasma nitrate and nitrite at 4 weeks of the LO-NI intervention
  Marker for nitrate bioavailability and functioning of the enterosalivary nitrate-nitrite-nitric oxide (NO) pathway
Change in blood monocyte-platelet aggregation | Change from baseline blood monocyte-platelet aggregation at 4 weeks of the HI-NI intervention
  Vascular inflammation biomarker
Change in blood monocyte-platelet aggregation | Change from baseline blood monocyte-platelet aggregation at 4 weeks of the LO-NI intervention
  Vascular inflammation biomarker
Change in high-sensitive plasma C-reactive protein (hsCRP) | Change from baseline plasma hsCRP at 4 weeks of the HI-NI intervention
  Inflammation biomarker
Change in high-sensitive plasma C-reactive protein (hsCRP) | Change from baseline plasma hsCRP at 4 weeks of the LO-NI intervention
  Inflammation biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Neubauer, Dr PhD, PD, Principal Investigator — University of Vienna
Locations (2):
- Austria (2):
  - Medical University of Vienna, Vienna
  - University of Vienna, Vienna

IPD SHARING:
Plan to Share IPD: Yes
For long-time preservation and sharing of the research data, it is planned to use the PHAIDRA digital repository of the University of Vienna (https://phaidra.univie.ac.at). This repository enables the permanent secure storage of digital assists including open access publications and research data necessary to reproduce and to verify the results of the publications.
  For all publications and other data related to this research that will be made available, all of the individual participant data collected during the trial will be de-identified.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The plan is to publish the findings in scientific journals and to present them at scientific meetings and to the public after the study is completed.
Access Criteria: Supporting the Open Access Policy of the University of Vienna, the PHAIDRA repository enables public access of the research data necessary to reproduce and to verify the results of publications from this research.

REFERENCES:
- [Background] Raubenheimer K, Hickey D, Leveritt M, Fassett R, Ortiz de Zevallos Munoz J, Allen JD, Briskey D, Parker TJ, Kerr G, Peake JM, Pecheniuk NM, Neubauer O. Acute Effects of Nitrate-Rich Beetroot Juice on Blood Pressure, Hemostasis and Vascular Inflammation Markers in Healthy Older Adults: A Randomized, Placebo-Controlled Crossover Study. Nutrients. 2017 Nov 22;9(11):1270. doi: 10.3390/nu9111270. PMID 29165355
- [Background] Raubenheimer K, Bondonno C, Blekkenhorst L, Wagner KH, Peake JM, Neubauer O. Effects of dietary nitrate on inflammation and immune function, and implications for cardiovascular health. Nutr Rev. 2019 Aug 1;77(8):584-599. doi: 10.1093/nutrit/nuz025. PMID 31150091
- [Background] Blekkenhorst LC, Bondonno NP, Liu AH, Ward NC, Prince RL, Lewis JR, Devine A, Croft KD, Hodgson JM, Bondonno CP. Nitrate, the oral microbiome, and cardiovascular health: a systematic literature review of human and animal studies. Am J Clin Nutr. 2018 Apr 1;107(4):504-522. doi: 10.1093/ajcn/nqx046. PMID 29635489
- [Derived] Fejes R, Pilat N, Lutnik M, Weisshaar S, Weijler AM, Kruger K, Draxler A, Bragagna L, Peake JM, Woodman RJ, Croft KD, Bondonno CP, Hodgson JM, Wagner KH, Wolzt M, Neubauer O. Effects of increased nitrate intake from beetroot juice on blood markers of oxidative stress and inflammation in older adults with hypertension. Free Radic Biol Med. 2024 Sep;222:519-530. doi: 10.1016/j.freeradbiomed.2024.07.004. Epub 2024 Jul 5. PMID 38972612
- [Derived] Fejes R, Lutnik M, Weisshaar S, Pilat N, Wagner KH, Stuger HP, Peake JM, Woodman RJ, Croft KD, Bondonno CP, Hodgson JM, Wolzt M, Neubauer O. Increased nitrate intake from beetroot juice over 4 weeks affects nitrate metabolism, but not vascular function or blood pressure in older adults with hypertension. Food Funct. 2024 Apr 22;15(8):4065-4078. doi: 10.1039/d3fo03749e. PMID 38546454